CLINICAL TRIAL: NCT03674437
Title: Evaluation of an Online, Remote Cognitive Battery for Use in Cancer Survivorship
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Dr. Susan Love Research Foundation (Other); ENFORMIA INC. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18-294
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Survivors
Keywords: Quality of Life; Cognitive Function; 18-294

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast Cancer Survivors: Each main cohort has 2 sub-groups: One sub-group in each main cohort will complete the traditional neurocognitive assessments and the Cogsuite Assessment at the MSK Counseling Center, and the other sub-group will complete the Cogsuite Assessment off-site, on their own computers, in a quiet space that is free of distractions.
  Interventions: Behavioral: Traditional Neurocognitive Assessments; Behavioral: Online Cognitive Battery (Cogsuite)
- Healthy Controls: Each main cohort has 2 sub-groups: One sub-group in each main cohort will complete the traditional neurocognitive assessments and the Cogsuite Assessment at the MSK Counseling Center, and the other sub-group will complete the Cogsuite Assessment off-site, on their own computers, in a quiet space that is free of distractions.
  Interventions: Behavioral: Traditional Neurocognitive Assessments; Behavioral: Online Cognitive Battery (Cogsuite)
- Healthy 21-25 year olds: Healthy participants between the ages of 21 and 25 will be administered the Cogsuite Battery remotely. These participants will not be matched to any other groups and will not be asked for their full medical histories. They will only complete the assessment only once.
  Interventions: Behavioral: Traditional Neurocognitive Assessments; Behavioral: Online Cognitive Battery (Cogsuite)

INTERVENTIONS:
Behavioral: Traditional Neurocognitive Assessments — Traditional Neurocognitive Assessments given with pen and paper
Behavioral: Online Cognitive Battery (Cogsuite) — Cognition (Cogsuite) for a battery that consists of seven measurements.

SUMMARY:
The purpose of this study is to measure changes in cognitive (mental) function in cancer survivors using a brief, reliable, game-like set of tests that can be completed outside the clinic, as an alternative to traditional neurocognitive assessments. This set of computerized tests, the Cogsuite Assessment, is expected to improve our ability to identify cognitive impairments in people who have been treated for cancer, so that we can (1) learn more about which cognitive functions are affected by cancer treatment, and (2) guide that treatment more effectively.

ELIGIBILITY:
Inclusion Criteria:

For All Participants:

* As per medical record or self-report,Female
* As per medical record or self-report,Age 40-65 at time of assessment
* Score of < 11 on the Blessed Orientation-Memory-Concentration Test (BOMC)
* As per self-report, If currently taking psychoactive medications (excluding gabapentin and including but not limited to antidepressants, and anxiolytics), on a daily basis dose must have been stable for at least two months prior to enrollment.
* English fluent (as per self-reported fluency of "very well")** ** Language verification: For both patients and controls, prior to enrollment, all will be asked the following two questions by an CRC to verify English fluency necessary for participation in the study:

  1. How well do you speak English? (must respond "Very well" when given the choices of Very well, Well, Not well, Not at all, Don"t know, or Refused)
  2. What is your preferred language for healthcare? (must respond English)

For Patients:

* As per medical record or self-report, female
* As per medical record or self-report, age 40-65 at time of assessment
* As per medical record or self-report, history of AJCC stages 0-3 breast cancer
* As per medical record or self-report, greater than six months post-treatment and within 10 years of treatment completion (Note: "post-treatment" refers to completion of surgery, radiation, and/or chemotherapy; a patient who is post-treatment but is on endocrine therapy is still eligible to participate.)

For Healthy Controls:

* As per medical record or self-report, female
* As per medical record or self-report, age 40-65 at time of assessment
* As per self-report, no history of cancer except non-melanoma/basal cell skin cancer/squamous cell skin carcinoma, and at the discretion of the PI, early stage secondary cancer diagnoses treated only with surgery (for example, endometrial or cervical cancer)

For Healthy 21-25 year old Group:

* As per medical record or self-report, age 21-25 at time of assessment
* As per self-report, no history of cancer except non-melanoma/basal cell skin cancer/squamous cell skin carcinoma, and at the discretion of the PI, early stage secondary cancer diagnoses treated only with surgery (for example, endometrial or cervical cancer)

Exclusion Criteria:

For All Participants:

* As per medical record or self-report, diagnosis of neurodegenerative disorder that affects cognitive function (e.g. Alzheimer"s disease, Parkinson"s disease, Multiple Sclerosis, Dementia, Seizure Disorders, etc.).
* As per medical record or self-report, history of stroke or head injury resulting in a structural lesion on neuropsych imaging, persistent cognitive difficulties impacting work or daily life or required cognitive rehabilitation.
* As per self-report, fine motor/motor impairments that interfere with participant"s ability to use a keyboard.
* As per medical record or self-report, a diagnosis of a Schizophrenia Spectrum Disorder, substance use disorder, Bipolar Disorder or Schizotypal personality disorder. Schizophrenia Spectrum Disorders include Schizophrenia, Schizophreniform disorder, Schizoaffective disorder, Delusional disorder, Brief psychotic disorder, and Attenuated Psychotic Disorder.
* As per medical record or self-report, visual or auditory impairment that would preclude ability to complete the assessments (e.g. history of significant macular degeneration or being unable to correct hearing with hearing aids)
* As per self-report, use of methotrexate (Amethopterin, Rhematrex, Trexall) or rituximab (Rituxan) for rheumatoid arthritis, psoriasis or Crohn"s disease, or cyclophosphamide (Cytoxan, Neosar) for Lupus.

For Patients only:

* As per medical record or self-report, history of another type of cancer, except non-melanoma/basal cell skin cancer/squamous cell skin carcinoma and, at the discretion of the PI, early stage secondary cancer diagnoses treated only with surgery (for example, endometrial or cervical cancer)

For all remote administrations:

* Minimum Hardware/Software Requirements*:

  * Processor: Intel Core i3 Processer or greater
  * Memory: 4GB RAM or greater
  * Operating System: Recent version of Windows or OS X
  * Browser: Google Chrome version 64 or higher
  * Internet Speed: 1.5 Mbps recommended
* As per self-report, a quiet space (home or office, door closed) to complete the assessments

  * Enformia Cognition will provide a web URL (https://www.cogsuite.com/testme) that participants can use to check if they have the minimum requirements. The URL will clearly state if the user has adequate hardware using green and red text and symbols. The test URL will also return a short 5 sequence numeric validation code (xx-xxx) for each browser checked. The validation code will allow Enformia to lookup the specific hardware that was tested. Research Associates can direct prospects to the test web URL during their phone screen.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer survivors
Study Population: MSK patients will be recruited through the survivorship clinics after having been identified via a Dataline query and/or weekly clinic schedules or through direct referrals from a member of the patient"s treatment team.
Sampling Method: Non-Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
validate computerized cognitive measures (Cogsuite Battery) | 2 years
  These will include 14 correlations, across the two cohorts and 7 tests (Modified Attention Network Test, N-Back Test, Stop-signal Test, Mental Rotation Test, Verbal Fluency Test, Motor Function Test, and Processing Speed Test).

CONTACTS AND LOCATIONS:
Overall Officials: James Root, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm